CLINICAL TRIAL: NCT05763810
Title: Analgesic Effects of Erector Spinae Plane Block Versus Superficial Parasternal Intercostal Plane Block Combined With Rectus Sheath Block After Off Pump Cardiac Surgery: A Randomised Trial
Brief Title: Comparing Different Regional Blocks for Analgesia After Off-pump Cardiac Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abd-Elazeem Abd-Elhameed Elbakry (Other)
Responsible Party: Sponsor-Investigator, Abd-Elazeem Abd-Elhameed Elbakry, Professor, Menoufia University
Organization: Menoufia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2/2023 ANET 15-3
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block group (Other): Erector Spinae Plane Block
  Interventions: Other: Erector Spinae Plane Block
- Superficial Parasternal Intercostal Plane Block and Rectus Sheath Block group (Other): Superficial Parasternal Intercostal Plane Block and Rectus Sheath Block
  Interventions: Other: Superficial Parasternal Intercostal Plane Block combined with Rectus Sheath Block

INTERVENTIONS:
Other: Erector Spinae Plane Block — Erector Spinae Plane Block
  Arms: Erector Spinae Plane Block group
Other: Superficial Parasternal Intercostal Plane Block combined with Rectus Sheath Block — Superficial Parasternal Intercostal Plane Block combined with Rectus Sheath Block
  Arms: Superficial Parasternal Intercostal Plane Block and Rectus Sheath Block group

SUMMARY:
This study aims to compare the analgesic effects of erector spinae plane block versus Superficial Parasternal Intercostal Plane Block block along with rectus sheath block after off-pump cardiac surgery

DETAILED DESCRIPTION:
General anaesthesia will be used for all patients. induction by midazolam 0.05-0.1 mg/kg, fentanyl 2-5 µ/kg, propofol 1-2 mg/kg, and atracurium 0.5 mg/kg for intubation. Maintenance by sevoflurane in oxygen-air mixture. regional blocks will be used after the induction of anaesthesia. Intraoperative analgesia will be maintained by fentanyl infusion 1-2 µ/kg/h while morphine sulphate 2.5-5mg will be used as rescue analgesia when pain score>4 beside acetaminophen 1000 mg /6 hours

ELIGIBILITY:
Inclusion Criteria:

* American Society of anaesthesiologists physical status classification II-III
* Elective off-pump cardiac surgery

Exclusion Criteria:

* Cognitive impairment
* Allergy to local anaesthetics
* Renal and/or hepatic dysfunction
* Ejection fraction< 45%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | Perioperative.
  µg and mg

SECONDARY OUTCOMES:
Pain intensity at rest and exercise | Perioperative.
  Visual analogue score: a score from 0 to 10(0= no pain and 10 the worst imaginable pain)
Extubation time | Perioperative
  minutes
Duration of post anaesthesia care unit stay | Perioperative
  minutes
Postoperative nausea | Perioperative
  number (%)
Postoperative vomiting | Perioperative
  number (%)
Duration of hospital stay | Postoperative up to 4 weeks
  days

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elazeem A Elbakry, MD, Principal Investigator — Menoufia University; Amal G Safan, MD, Principal Investigator — Menoufia University; Islam M El-Desoky, MD, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Medicine, Cairo, Shebin Elkom, Egypt